CLINICAL TRIAL: NCT04873804
Title: The Effect Of Transcranial Direct Stimulation Applied To The Dorsolateral Prefrontal Cortex And Posterior Parietal Cortex İn Cognitive Function, Mood And Proprioception İn Healthy Adults
Brief Title: The Effect of Transcranial Direct Stimulation on Cognitive Functions of Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Damla Ören, Physiotherapist MSc, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: tDCS on DLPFC and PPC
Record Dates: First submitted 2021-04-14; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Symptom; Healthy
Keywords: tDCS; Dorsolateral Prefrontal Cortex; Posterior Parietal Cortex; Cognitive Function
MeSH Terms: conditions — Neurobehavioral Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LEFT DLPFC (Active Comparator): The anode electrode of tDCS was applied to the left DLPFC and the cathode electrode was connected to the contralateral shoulder.
  Interventions: Other: Transcranial Direct Current Stimulation
- RİGHT PPC (Active Comparator): The anode electrode of tDCS was applied to the right PPC and the cathode electrode was connected to the contralateral shoulder.
  Interventions: Other: Transcranial Direct Current Stimulation
- Sham (Sham Comparator): Placebo was applied by placing the electrodes in the right PPC and left DLPFC without applying current.
  Interventions: Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — The intervention protocols were applied using tDCS (Teknofil TESsaNova). All individuals received 2 mA of anodal tDCS for 2 weeks on weekdays. All applications were done in the form of 20-minute sessions.

SUMMARY:
Background: Transcranial direct current stimulation(tDCS) has been used to improve cognitive functions in healthy young adults.

Purpose: To investigate the effect of TDCS application on different cortex regions on cognitive function.

Methods: Sixty individuals aged 18-30 were included in the study. The participants were randomly divided into the left dorsolateral prefrontal cortex (Left DLPFC Group)(n=20), the right posterior parietal cortex (Right PPC Group)(n=20), and the sham group (Sham Group)(n=20). tDCS was applied for 20 minutes on weekdays for 2 weeks. The participants were evaluated in terms of cognitive functions with Neuropsychometric Test Battery before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* being 18-30 years old

Exclusion Criteria:

* alcohol and substance addiction
* previous mental illness
* having mental and cognitive problems
* a history of head trauma
* having cardiovascular disease.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Test Battery | 3 weeks
  It is a test battery for getting detailed information about general cognitive status.
Beck Depression Scale | 3 weeks
  It measures the symptoms seen in depression such as emotional, cognitive and motivational. It includes 21 items determine a behavioral feature related to depression. Items are numbered from 0 to 3. The goal is to objectively break down the degree of symptoms.
  The total score of all answers is calculated as follows:
  0 to 9 points: Minimally depressive symptoms 10 to 16 points: Mild depressive symptoms Between 17 and 29 points: Moderate depressive symptoms Between 30 and 63 points: Severe depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Miray Budak, PhD, Principal Investigator — Medipol University; Lutfu Hanoglu, PhD, Study Chair — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Damla Ören, Istanbul
  - Medipol Mega Hospital, Istanbul